CLINICAL TRIAL: NCT00751166
Title: A Comparative Double-blind, Double-dummy Study of Desloratadine (DL) 5 mg Once Daily, Cetirizine 10 mg Once Daily, and Placebo Once Daily in Patients With Chronic Idiopathic Urticaria (CIU)
Brief Title: A Comparative Double-blind, Double-dummy Study of Desloratadine (DL) 5 mg Once Daily, Cetirizine 10 mg Once Daily, and Placebo Once Daily in Patients With Chronic Idiopathic Urticaria (Study P03736)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study could not be re-supplied with study medication in a timely manner.
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P03736
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Urticaria
MeSH Terms: conditions — Urticaria | interventions — desloratadine; Cetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Desloratadine
  Interventions: Drug: Desloratadine
- 2 (Active Comparator): Cetirizine
  Interventions: Drug: Cetirizine
- 3 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Desloratadine — Desloratadine 5 mg, oral tablet, once daily in the morning, 28 days
  Arms: 1
Drug: Cetirizine — Cetirizine 10 mg, oral tablet (over encapsulated), once daily in the morning, 28 days
  Arms: 2
Drug: placebo — placebo once daily for 28 days
  Arms: 3

SUMMARY:
This was a randomized, double-blind, parallel-group, multicenter study that used both an active control (cetirizine) and a placebo control to evaluate desloratadine 5 mg once daily during a 28-day treatment period. The active treatments and placebo were allocated in a 2:2:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Have demonstrated their willingness to participate in the study and comply with its procedures by signing a written informed consent. For pediatric patients, the parent or legal guardian was to have signed a written informed consent.
* Be between 12 and 70 years of age, of either sex and any race.
* Have had signs and symptoms of CIU for at least 6 weeks prior to the Screening Visit.
* Have been experiencing a current flare of their CIU of at least 3 weeks prior to the Baseline Visit. Hives were to have been present for at least 3 days per week during the current flare prior to the Baseline Visit.
* Have an overall condition of CIU that was at least of "moderate" severity (minimum score of 2) at both Screening and Baseline Visits.
* Have at least a moderately severe pruritus score (minimum score of 2) and hives (minimum score of 1) present at Screening.
* Have, at Baseline, a total pruritus score of 14 or greater for the sum of AM and PM (reflective) diary scores for the 3 days prior to Baseline and the AM diary score on Day 1.
* Understand and be able to adhere to the dosing and visit schedules, and agree to assess and record their symptom severity scores, medication times,concomitant medications, and adverse events accurately and consistently in a daily diary.
* Be in general good health and free of any clinically significant disease (other than CIU) that would have interfered with study evaluations.
* If female and of childbearing potential, have had a negative urine (hCG) pregnancy test at the time of Baseline (Visit 2).
* Female subjects of childbearing potential were to be counseled in the appropriate use of birth control while in the study. They were to be using a medically accepted method of birth control, for example: double barrier method, oral contraceptive, Depo-Provera®, or Norplant®, prior to Baseline and during the study. Women who were not sexually active were to agree and consent to use one of the above-mentioned methods should they become sexually active while participating in the study. If the subject had had a tubal ligation or was using an intra-uterine device, or if the husband/partner had had a vasectomy, another method was to be used.

Exclusion Criteria:

* Had asthma requiring chronic use of inhaled or systemic corticosteroids.
* Had been unresponsive to antihistamine treatment in the past.
* Had a history of allergies to more than two classes of medication or who were allergic to or unable to tolerate antihistamines.
* Had used any investigational drug in the last 30 days prior to Baseline.
* Had food or drug allergies manifested as skin reactions. Subjects with urticaria that was primarily due to physical urticaria or other known etiology.
* If female, were pregnant or nursing.
* Had a history of hypersensitivity to the study drug or its excipients.
* Were family members of the investigational study staff involved with this study.
* Had previously been randomized into the study.
* Had current evidence of clinically significant hematopoietic, cardi distribution, metabolism, or excretion of the study medication or with the subject's ability to reliably complete the diary card.
* Were morbidly obese (BMI >= 35, as described in Appendix 6 of the protocol)
* Had a compromised ability to provide informed consent.
* Had a history of non-compliance with medications or treatment protocols.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2004-03-01 (Actual); Primary Completion 2005-05-01 (Actual); Study Completion 2005-05-01 (Actual)

PRIMARY OUTCOMES:
Compare the efficacy of the study treatments with respect to the change from Baseline in the average AM/PM 12-hour reflective pruritus severity score (diary recordings) | After the first 7 days of treatment

SECONDARY OUTCOMES:
Joint physician-patient evaluations ("now") of: overall condition of the CIU and overall global therapeutic response. | At treatment days 14 and 28 (Visit 3 and 4)
Average AM/PM "reflective" diary scores over treatment days 1-7, 8-14, 15-21 and 22-28 for: severity of pruritus; number of hives; size of largest hives; total symptom score (pruritus, number of hives, size of the largest hives) | Days 7, 14, 21 and 28
Average AM/PM "reflective" diary scores over treatment days 1-7, 8-14, 15-21 and 22-28 for: subject-evaluated CIU interference with sleep (AM) and interference with daily activities (PM) | Days 7, 14, 21 and 28
Adverse Events | End of Trial